CLINICAL TRIAL: NCT06189573
Title: Reconstruction of the Anterior Cruciated Ligament With Quadriceps Tendon Graft With Bone Plug vs Bone Patellar Tendon Bone Graft, a Randomized Clinical Controlled Essay With 2 Years of Follow up
Brief Title: Reconstruction of the ACL With QT Graft With Bone Plug vs BPTB
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Responsible Party: Principal Investigator, Dr. Félix Enrique Villalobos Córdova, MD PhD, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Por asignar
Record Dates: First submitted 2023-12-02; First posted 2024-01-03 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior Cruciate Ligament Reconstruction; Bone patellar tendon bone graft; Quadriceps tendon graft; KT-1000; IKDC
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Intervention Model Description: Controlled, longitudinal, prospective, randomized, double-blind clinical trial that will include patients from the Luis Guillermo Ibarra-Ibarra National Rehabilitation Institute (INRLGII) of the Sports Orthopedics and Arthroscopy service, with primary ACL injury who undergo surgery with a consistent procedure in ACL reconstruction either with the use of bone tendon bone graft or quadriceps tendon with bone pad in the period from October 2023 to October 2025.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The selection of the graft to be used will be carried out randomly with a box with a closed envelope, which contains the same number of envelopes with one or another type of graft, and the resulting option will be the way in which the type of graft is assigned. graft, which will not be disclosed to the patient during the period of the study.
  Subjective and objective clinical evaluations with KT-1000 will be carried out preoperatively and postoperatively at 3, 6, 12 and 24 months by 2 evaluators who will be blinded to the type of graft used in each patient, for which the anterior part of his knee will be covered with a 20cm long "micropore" band, so that the type of graft cannot be identified by the evaluator based on the area of the knee and surgical scar.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quadriceps Tendon graft (Other): Patients with ACL reconstruction with the use of quadriceps tendon graft
  Interventions: Procedure: Anterior cruciate ligament Reconstruction with autologous quadriceps tendon graft
- Bone Patellar Tendon Bone Graft (Other): Patients with ACL reconstruction with the use of bone patellar tendon bone graft
  Interventions: Procedure: Anterior cruciate ligament Reconstruction with autologous bone patellar tendon bone graft

INTERVENTIONS:
Procedure: Anterior cruciate ligament Reconstruction with autologous quadriceps tendon graft — Surgical reconstruction of anterior cruciate ligament with autologous quadriceps tendon graft
  Arms: Quadriceps Tendon graft
Procedure: Anterior cruciate ligament Reconstruction with autologous bone patellar tendon bone graft — Surgical reconstruction of anterior cruciate ligament with autologous bone patellar tendon bone graft
  Arms: Bone Patellar Tendon Bone Graft

SUMMARY:
Background: Anterior cruciate ligament (ACL) injury is one of the most common orthopedic injuries worldwide. Currently, the use of the bone patellar tendon bone graft (BPTB) technique is considered the gold standard. The use of the quadriceps tendon graft (QT) has gained greater interest in recent years, this because with an adequate technique it is possible to obtain a biomechanically superior graft with fewer adverse events. The objective of this study is to compare the objective and subjective clinical results, as well as the presence or not of adverse events in ACL reconstruction with these 2 types of grafts in the medium term.

Materials and methods: Controlled, longitudinal, prospective, randomized, double-blind clinical trial that will include patients of both sexes, between 15 and 55 years of age, with primary ACL injury who attend the outpatient clinic of the Sports Orthopedics Service. INRLGII arthroscopy between October 2023 and October 2025, prior informed consent. Graft selection will be done randomly 1:1 between bone-tendon-bone (BPTB) graft Vs. quadriceps tendon graft (QT) for ACL reconstruction surgery. The clinical evaluation of the patients Will be done by 2 blinded evaluators, through the objective measurement of KT-1000 and the use of subjective clinical knee scales, both preoperatively and at 3-6-12 and 24 months. The presence or absence of adverse events or complications will be documented during a minimum of 2 years of follow-up. Parametric and non-parametric statistical tests will be used depending on whether the distribution is normal or not, for dependent and independent groups, using the SPSS version 25 statistical program.

DETAILED DESCRIPTION:
JUSTIFICATION ACL rupture is one of the most frequent and studied injuries in orthopedic literature. Various short-, medium- and long-term results of ACL reconstruction have been described in the international literature, as well as comparisons between different types of reconstruction techniques, grafts and complications.

The vast majority of studies and clinical trials focus on BPTB and hamstrings tendon (HT), the former being considered by multiple authors as the gold standard for the management of these injuries despite its association with high donor site morbidity such as anterior knee pain, pain when kneeling and muscle weakness.

With an adequate surgical technique for both graft harvesting and ACL reconstruction, the use of QT as a graft has reported good biomechanical and clinical results and even superior to other grafts. However, despite this, at present a precise justification has not been established that defines the advantages or disadvantages of choosing this graft over other popular techniques, which is why a randomized study was carried out in a center of high specialty and concentration of patients with this type of lesions will increase the level of scientific validation of the information available regarding the use of this graft.

PROBLEM STATEMENT Is there a statistically significant difference between both techniques (BPTB and QT) at 2 years? Minimum follow-up regarding clinical evolution measured with IKDC, objective stability measured by KT-1000, and adverse events in primary ACL reconstruction?

HYPOTHESIS In patients with anterior cruciate ligament (ACL) injury who undergo surgery reconstruction with the use of autologous quadriceps tendon with bone plug (QT) or bone patellar tendon bone (BPTB) graft, there will be no statistically significant difference between them, in the first 2 years of follow-up, in terms of clinical evolution measured by the International subjective scale Knee Documentation Committee (IKDC), nor objective stability measured by arthrometry with the KT1000 device; In addition, there will be fewer adverse events in patients in whom quadriceps tendon graft (QT) was used compared to bone patellar tendon bone graft (BPTB).

GENERAL OBJECTIVE Observe if there is a statistically significant difference between both QT and BPTB grafts in terms of clinical evolution measured by IKDC, and objective stability measured by KT-1000, as well as reporting adverse events in both groups at 2 years of follow-up.

MATERIAL AND METHODS Controlled, longitudinal, prospective, randomized, double-blind clinical trial that will include patients from the Luis Guillermo Ibarra-Ibarra National Rehabilitation Institute (INRLGII) of the Sports Orthopedics and Arthroscopy service, with primary ACL injury who undergo surgery with a consistent procedure in ACL reconstruction either with the use of bone patellar tendon bone graft or quadriceps tendon with bone pad in the period from October 2023 to October 2025. When a patient who requires ACL reconstruction surgery is scheduled in our service, if he meets With the inclusion criteria, you will be invited to participate in the study and if you accept and give your written informed consent you will be included in the study. The selection of the graft to be used will be carried out randomly with a box with a closed envelope, which contains the same number of envelopes with one or another type of graft, and the resulting option will be the way in which the type of graft is assigned. graft, which will not be disclosed to the patient during the period of the study. During the surgical procedure, the repair of concomitant injuries (meniscal or chondral) will be carried out, and at the end of the surgery, the surgeon will prepare the surgical report sheet detailing the findings found and the characteristics of the graft used in terms of thickness, length , and the presence or absence of incidents during surgery.

Subjective clinical scales from IKDC, Kujala, Lysholm, Tegner, and KOOS will be applied. Measurement of the anterior translation of the tibia will be performed objectively with the use of the KT-1000 device.

Subjective and objective clinical evaluations with KT-1000 will be carried out preoperatively and postoperatively at 3, 6, 12 and 24 months by 2 evaluators who will be blinded to the type of graft used in each patient, for which the anterior part of his knee will be covered with a 20cm long "micropore" band, so that the type of graft cannot be identified by the evaluator based on the area of the knee and surgical scar. Clinical follow-up of the patient will also be carried out, in the necessary weeks or months at the discretion of the surgeon or treating doctor, as is usually carried out in the clinical practice of the institute.

Non-contrast magnetic resonance imaging (MRI) studies will be performed to evaluate the integrity of the ACL graft, by an orthopedic evaluator with experience in musculoskeletal imaging, blinded to the type of graft used, to classify it as: intact graft, graft with partial injury to its fibers or graft with complete injury to its fibers. Knee radiographs will also be performed (AP projection in standing position, lateral at 30° of flexion and axial of the patella at 40°), preoperatively and 12 and 24 months after surgery, which will be evaluated by an orthopedic evaluator with experience in musculoskeletal imaging. , blinded to the type of graft used, to evaluate the presence or absence of Osteoarthritis according to the Kellgren & Lawrence classification, in grades 0 to 4.

All patients will be subjected to the same rehabilitation protocol during the first 3-4 months after surgery, as well as follow-up by sports medicine both pre-surgery and from the 3rd to 4th post-surgical month to receive the same muscle strengthening protocol established in our Institute for patients undergoing ACL reconstruction surgery. Keeping a record of the evaluation of preoperative and postoperative quadriceps strength in a standardized and objective manner through isokinetic evaluation with Cybex.

The use of a mechanical knee brace locked to the operated on knee will not be required on a routine basis, unless there is some indication of its use by the treating surgeon to protect associated injuries that require it, and in that case the use of It will be for a period of no more than 6 weeks. Patients must perform assisted ambulation with the use of crutches for the first 2 weeks with partial support of the operated leg and will subsequently progress to full support, as long as there is no contraindication on the part of the treating surgeon in relation to the management of associated injuries.

The presence or absence of adverse events or complications will be documented during 2 years of minimal monitoring. Parametric and non-parametric statistical tests will be used depending on whether the case has a normal distribution or not, for dependent and independent groups, of the related variables that are the result of periodic evaluations (3, 6, 12 and 24 months) of the same technique. either QT or BPTB, using the SPSS statistical program version 25.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 15 to 55 years old.
* Primary ACL rupture diagnosed by MRI.
* INR-LGII patients with a complete institutional record.
* Without the presence of systemic, chronic degenerative comorbidities that could affect the quality of the graft. (Diabetes, Thyroid, Autoimmune diseases).

Exclusion Criteria:

* Grade 2 or 3 posterior cruciate ligament injuries.
* Multiligamentous injuries.
* Severe varus/valgus deformities (mechanical axis outside the range of 35% to 65% of the articular surface of the tibia).
* Previous knee surgeries to be treated.
* Anterior knee pain present (VAS greater than 6), with brush and escape maneuvers positive.
* K&L osteoarthritis ≥ 2 in the knee to be treated.
* History of intra-articular fractures of the injured knee.
* History of ACL injury and/or surgery in the contralateral knee.
* Previous injury to the patellar or quadriceps tendon (total or partial rupture).
* Symptomatic extensor mechanism tendinopathies.
* High patella (Caton-Deschamps index 1.2 mm)
* ICRS grade III or IV chondral lesion in patella greater than 1cm 2
* Medical conditions that prevent full patient participation (e.g. cancer active, rheumatoid arthritis, etc.)
* Pregnancy.
* Obesity (WCC >30).

Perioperative elimination criteria:

* Medial or lateral meniscus injury >50% non-repairable.
* Medial and/or lateral menisectomy > 50%
* Grade 2-3 ligament instability associated with ACL injury.
* Cartilage lesion >2 cm2 ICRS grade 3-4, untreated.
* Associated surgeries due to instability.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee score (IKDC) | Presurgical, 3, 6, 12 and 24 postsurgical months
  Minimum value 0 Maximum value 100 Higher scores mean a better outcome Subjective assesment. Three categories are examined by the questionnaire: symptoms, athletic activity, and knee function
KT-1000 | Presurgical, 3, 6, 12 and 24 postsurgical months
  Device for objective stability measurement.

SECONDARY OUTCOMES:
Anterior Knee Pain Scale (Kujala score) | Presurgical, 3, 6, 12 and 24 postsurgical months
  Minimum value 0 Maximum value 100 Higher scores mean a better outcome Subjective assesment for anterior knee pain
Lysholm Knee Scoring Scale | Presurgical, 3, 6, 12 and 24 postsurgical months
  Minimum value 0 Maximum value 100 Higher scores mean a better outcome Subjective assesment for knee instability
Tegner Activity Scoring Scale | Presurgical, 3, 6, 12 and 24 postsurgical months
  Minimum value 0 Maximum value 10 Higher scores mean a better outcome Activity assesment
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Presurgical, 3, 6, 12 and 24 postsurgical months
  Minimum value 0 Maximum value 100 Higher scores mean a better outcome Subjective assesment for knee injuries

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Rehabilitacion Luis Guillermo Ibarra Ibarra, Mexico City, Mexico City, Mexico